CLINICAL TRIAL: NCT00087087
Title: A Phase II Evaluation Of Pemetrexed (ALIMTA LY231514, IND #40061) In The Treatment Of Recurrent Or Persistent Platinum-Resistant Ovarian Or Primary Peritoneal Carcinoma
Brief Title: Pemetrexed Disodium in Treating Patients With Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Masking: None | Purpose: Treatment
Other Study IDs: GOG-0126Q; LILLY-H3E-US-JMGP; CDR0000372919
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: pemetrexed disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pemetrexed disodium, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well pemetrexed disodium works in treating patients with recurrent or persistent ovarian epithelial cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of pemetrexed disodium in patients with recurrent or persistent platinum-resistant ovarian epithelial or primary peritoneal cancer that failed higher priority treatment protocols.
* Determine the nature and degree of toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Beginning 7 days before and continuing until 3 weeks after the last dose of pemetrexed disodium, patients also receive oral folic acid daily and cyanocobalamin (vitamin B_12) intramuscularly every 9 weeks.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 19-51 patients will be accrued for this study within 11-22 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial or primary peritoneal cancer

  * Recurrent or persistent disease
* Measurable disease

  * At least 1 unidimensionally measurable target lesion ≥ 20 mm by conventional techniques (e.g., palpation, plain x-ray, CT scan, or MRI) OR ≥ 10 mm by spiral CT scan
  * Tumors within a previously irradiated field are considered non-target lesions
* Must have received 1 prior platinum-based (carboplatin, cisplatin, or another organoplatinum compound) chemotherapy regimen for primary disease

  * Initial treatment may have included high-dose therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment
  * Patients who had not received prior paclitaxel may have received a second regimen that included paclitaxel
* Platinum-resistant or refractory disease

  * Treatment-free interval < 6 months after prior platinum-based therapy OR progressed during platinum-based therapy
* Not eligible for a higher priority GOG protocol (i.e., any active phase III GOG protocol for the same patient population)

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN*
* AST and ALT ≤ 3 times ULN* NOTE: * ≤ 5 times ULN if due to hepatic metastases

Renal

* Creatinine clearance ≥ 45 mL/min

Other

* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No neuropathy (sensory or motor) > grade 1
* No active infection requiring antibiotics
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* One prior noncytotoxic (biologic or cytostatic) regimen allowed for management of recurrent or refractory disease, including, but not limited to, the following:

  * Monoclonal antibodies
  * Cytokines
  * Small-molecule inhibitors of signal transduction
* At least 3 weeks since prior biologic or immunologic therapy
* At least 24 hours since prior growth factors
* No concurrent routine colony-stimulating factors

Chemotherapy

* See Disease Characteristics
* Recovered from prior chemotherapy
* No prior cytotoxic chemotherapy for recurrent or persistent disease, including retreatment with initial chemotherapy regimens
* No prior pemetrexed disodium

Endocrine therapy

* At least 1 week since prior hormonal therapy for the malignant tumor
* Concurrent hormone replacement therapy allowed

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy to > 25% of bone marrow
* At least 2 weeks since prior radiotherapy and recovered

Surgery

* Recovered from prior surgery

Other

* No prior cancer treatment that would preclude study participation
* No non-steroidal anti-inflammatory drugs (NSAIDs) for 2-5 days before, during, and for 1-2 days after study drug administration

  * Concurrent low-dose (≤ 325 mg/day) aspirin allowed
* At least 3 weeks since other prior therapy for the malignant tumor

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2004-07; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Antitumor activity
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: David S. Miller, MD, Study Chair — Simmons Cancer Center
Locations (35):
- United States (35):
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Women's Cancer Center - Las Vegas, Las Vegas, Nevada
  - UMDNJ University Hospital, Newark, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Care Associates - Midtown Tulsa, Tulsa, Oklahoma
  - Williamette Gynecologic Oncology PC, Salem, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Baptist Regional Cancer Center at Baptist Hospital of East Tennessee, Knoxville, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia